CLINICAL TRIAL: NCT02871297
Title: Long-term, Open-label, Flexible-dose, Extension Study of Vortioxetine in Child and Adolescent Patients With Major Depressive Disorder (MDD) From 7 to 18 Years of Age
Brief Title: Long-term, Open-label, Flexible-dose, Extension Study of Vortioxetine in Child and Adolescent Participants With Major Depressive Disorder (MDD) From 7 to 18 Years of Age
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated based on new efficacy data from another study.
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12712A; 2008-005356-25 (EudraCT Number)
Record Dates: First submitted 2016-08-15; First posted 2016-08-18 (Estimated); Results first posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-11

CONDITIONS: Depressive Disorder, Major
Keywords: adolescent; children
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vortioxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vortioxetine (Experimental): Vortioxetine tablets for 26 weeks. Single dose of vortioxetine oral drops (only a subset of participants).
  Interventions: Drug: Vortioxetine

INTERVENTIONS:
Drug: Vortioxetine — Target dose is 10 mg/day, however, the dose can be down- or uptitrated to 5, 15, or 20 mg/day.
  Other Names: Brintellix (R); Lu AA21004

SUMMARY:
Evaluation of the long-term safety and tolerability of vortioxetine in child and adolescent participants with a Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5™) diagnosis of MDD.

ELIGIBILITY:
Inclusion Criteria:

* The participant is a male or female child aged ≥7 and <12 years or adolescent aged ≥12 and ≤18 years in the lead-in study (12709A and 12710A).
* The participant must have completed Study 12709A or 12710A (Visit 12, Completion Visit) immediately prior to enrolment into this extension study.
* The participant had a primary diagnosis of MDD at entry in study 12709A or 12710A, diagnosed according to DSM-5™.
* The participant is indicated for long-term treatment with vortioxetine according to the clinical opinion of the Investigator.
* For participants aged ≥7 and ≤17 years at the Baseline visit; the participant is able to understand the Informed Assent Form, and parent(s)/legal representative(s) are able to read and understand the Informed Consent Form.
* For participants who turned 18 years during the lead-in study 12710A; the participant has signed the Informed Consent Form.

Exclusion Criteria:

* The participant has been diagnosed with another psychiatric disorder (for example mania, bipolar disorder, schizophrenia or any psychotic disorder) during study 12709A or 12710A.
* The participant has an attention-deficit/hyperactivity disorder (ADHD) that requires a pharmacological treatment other than a stimulant medication.

Other protocol-defined inclusion and exclusion criteria may apply

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 662 (Actual)
Dates: Start 2016-08-17 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (78):
- United States (4):
  - The University of Arizona Sarver Heart Center (SHC), Tucson, Arizona
  - Kansas University School of Medicine-Wichita, Wichita, Kansas
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University Hospital Cleveland Medical Center Division of Child and Adolescent Psychiatry, Cleveland, Ohio
- Bulgaria (2):
  - MHAT Targovishte AD, Targovishte
  - Diagnostic Consultative Center Mladost-M Varna OOD, Varna
- Paediatric Sleep Research Inc., Toronto, Ontario, Canada
- Colombia (4):
  - E.S.E. Hospital Mental de Antioquia HOMO, Bello, Antioquia
  - Centro de Investigaciones y Proyectos en Neurociencias CIPNA LTDA IPS., Barranquilla, Atlántico
  - Centro de investigaciones del Sistema Nervioso SAS Grupo CISNE SAS, Bogotá, DC
  - Psynapsis Salud Mental S.A., Pereira, Risaralda Department
- Marienthali Kliinik, Tallinn, Estonia
- France (3):
  - Cabinet Psyche, Douai, Nord
  - Centre Medical Ambroise Pare, Élancourt
  - CHU de Nantes - Hopital Hotel Dieu, Nantes
- Germany (4):
  - Univ. Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Rheinhessen-Fachklinik Mainz, Kinder und Jugendpsychiatri, Mainz
  - Klinik fur Kinderneurologie und Sozialpadiatrie Kinderzentrum Maulbronn gGmbH, Maulbronn
  - University Hospital Tuebingen -, Tübingen
- Hungary (2):
  - Vadaskert Child Psychiatric Hospital and Outpatient, Budapest
  - Bekes Megyei Kozponti Korhaz Pandy Kalman Tagkorhaza, Gyula
- Ramat Chen - Mental Health Clinic, Tel Aviv, Israel
- Italy (6):
  - Scientific Institute Fondazione Stella Maris, Calambrone, Pisa
  - Sciaf Ulss 16 Padova, Padua, Regione Veneto
  - Hospital Trust-University of Cagliari, Cagliari
  - U.O.C. Neuropsichiatria Infantile - IRCCS Istituto Giannina Gaslini, Genova
  - Dip.Sc.Biomediche, Odont. e Imm.Funz.li, AOU Policlinico G. Martino, Messina
  - University Federico II Of Naples, Napoli
- Latvia (4):
  - Hospital Gintermuiza, Jelgava
  - Linda Keruze's Psychiatric Center, LLC, Liepāja
  - Children Hospilal -Gailezers, Riga
  - Sigulda Hospital Outpatient Clinic, Sigulda
- Mexico (7):
  - Clinica Cemelli, Guadalajara, Jalisco
  - Roberto Zepeda Sanchez, Guadalajara, Jalisco
  - Instituto Nacional de Pediatria (INP) (National Institute of Pediatrics), Mexico City, Mexico City
  - CRI Centro Regiomontano de Investigacion SC, Monterrey, Nuevo León
  - Centro para el Desarrollo de la Medicina y de Asistencia Medica Especializada S.C, Culiacan de Rosales, Sinaloa
  - B & B Investigaciones Medicas, SC, Mazatlán, Sinaloa
  - BIND Investigaciones S.C, San Luis Potosí City
- Poland (7):
  - Prywatne Gabinety Lekarskie Promedicus, Bialystok, Podlaskie Voivodeship
  - Centrum Badan Klinicznych PI-House Sp. z o.o., Gdansk
  - Przychodnia Syntonia Poradnia Zdrowia Psychicznego, Kielce
  - Spectrum Centrum Psychiatrii Specjalistyczny Gabinet Psychiatryczny, Lublin
  - Filip Rybakowski Specjalistyczna Praktyka Lekarska, Poznan
  - Specjalistyczny Szpital im. dra A. Sokolowskiego w Walbrzychu, Wałbrzych
  - Centrum Neuropsychiatrii Neuromed, Wroclaw
- Russia (15):
  - Medicorehabilitation Research Center Phoenix, Rostov-on-Don, Rostov State
  - Stavropol Region Psychiatric Hospital No.2, Stavropol, Stavropol Kray
  - Arkhangelsk Regional Clinical Mental Hospital, Arkhangelsk
  - GUZ Engels Psychiatric Hospital, Engel's
  - State Budgetary Healthcare Institution (SBHI) Specialized Clinical Psychiatric Hospital 1 of the ..., Krasnodar
  - Lipetsk Regional Psychoneurological Hospital, Lipetsk
  - Nizhny Novgorod Region State Institution Of Healthcare Clinical Psychiatric Hospital 1 Of Nizhny ..., Nizhny Novgorod
  - LLC City Neurological Center Sibneuromed, Novosibirsk
  - Rostov State Medical University of the Minzdravsotsrazvitiya of Russia, Rostov-on-Don
  - City Psychiatric Hospital No.3 named after I.I. Skvortsov-Stepanov, Saint Petersburg
  - Saratov State Medical University, Saratov
  - Guz Saratov Regional Psychiatric Hospital St. Sofii, Saratov
  - Nebbiolo LLC, Tomsk
  - Yaroslavl Regional Clinical Psychiatry Hospital, Yaroslavl
  - State Budgetary Healthcare Institution of Sverdlovsk Region Â¿Sverdlovsk Regional Clinical Psychi..., Yekaterinburg
- Serbia (5):
  - Child and Adolescent Neurology and Psychiatry Clinic, Belgrade
  - Institute of Mental Health, Belgrade
  - University Clinical Center Kragujevac, Kragujevac
  - Clinical Center of Vojvodina - Clinic of Psychiatry, Novi Sad
  - Daily Hospital for Children and Adolescents, Pantelej-Nis
- Cape Trial Centre, Bellville, Cape Town, South Africa
- South Korea (2):
  - Soon Chun Hyang University Hospital Cheonan, Cheonan-si, Chungcheongnam-do
  - Asan Medical Center, Seoul
- Spain (3):
  - Hospital Universitario Fundacion Alcorcon, Alcorcón, Madrid
  - Unidad de Salud Mental Infanto-Juvenil (USMI-J) Edificio de Consultas Externas. Hospital MarAtimo, Torremolinos, Malaga
  - Hospital General Universitario Gregorio Maranon, Madrid
- Ukraine (4):
  - Ukrainian Research Institute Of Social, Forensic Psychiatry And Drug Abuse, Kiev City Psychoneuro..., Kyiv
  - Odessa Regional Medical Centre of Mental Health, Odesa
  - Maltsev Poltava Regional Clinical Psychiatric Hospital, Higher State Educational Institution Of U..., Poltava
  - Ternopil Regional Clinical Municipal Psycho-Neurological Hospital, Ternopil State Medical Univers..., Ternopil
- United Kingdom (2):
  - NHS Greater Glasgow and Clyde Glasgow Clinical Research Facility-Queen Elizabeth University Hospi..., Glasgow
  - Alder Hey Hospital, Liverpool

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a long-term extension study in child and adolescent participants with MDD who completed 1 of the double-blind, placebo-controlled, active-reference Study 12709A (NCT02709655) or 12710A (NCT02709746).
Groups:
- Vortioxetine: Participants initiated treatment with vortioxetine 5 milligrams (mg)/day orally for the first 2 days and thereafter they received 10 mg/day vortioxetine. Based on the response and dose-limiting adverse events (AEs), vortioxetine dose could be up- or down-titrated with 5 mg/day but the maximum dose did not exceed 20 mg/day. The total duration of treatment was 26 weeks.
Period: Overall Study
Arm/Group | Vortioxetine
Started | 662
Received at Least 1 Dose of Study Drug | 662
Completed | 526
Not Completed | 136
Not completed — Adverse Event | 34
Not completed — Lack of Efficacy | 10
Not completed — Non-compliance with study drug | 15
Not completed — Protocol Violation | 3
Not completed — Withdrawal by Subject | 20
Not completed — Lost to Follow-up | 13
Not completed — Rolled over to 13546A | 2
Not completed — Other than specified | 39

BASELINE CHARACTERISTICS:
Population: All-patients-treated set (APTS) included all participants who took at least 1 dose of vortioxetine in this study 12712A.
Groups:
- Vortioxetine: Participants initiated treatment with vortioxetine 5 mg/day orally for the first 2 days and thereafter they received 10 mg/day vortioxetine. Based on the response and dose-limiting AEs, vortioxetine dose could be up- or down-titrated with 5 mg/day but the maximum dose did not exceed 20 mg/day. The total duration of treatment was 26 weeks.
Arm/Group | Vortioxetine
Number analyzed (Participants) | 662
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.33 (3.07) [lower limit 3.07]
Age, Customized [Count of Participants; unit: Participants]
  Children (7-11 years) | 300
  Adolescents (12-17 years) | 352
  Adults (18-64 years) | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 361
  Male | 301
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 447
  Black | 8
  Asian | 5
  Other | 188
  Unknown | 9
  Not reported | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. SAEs included death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized the participant and required medical intervention to prevent 1 of the outcomes listed in this definition. TEAE was defined as an AE that started or increased in intensity on or after the date of first dose of study drug in this study 12712A. A summary of serious and non-serious AEs regardless of causality is located in 'Reported Adverse Events module'.
Time Frame: Baseline up to Week 30
Population: APTS included all participants who took at least 1 dose of vortioxetine in this study 12712A.
Measure: Count of Participants; unit: Participants
Arm/Group | Vortioxetine
Number analyzed (Participants) | 662
Participants | 404

2. Secondary Outcome: Change From Baseline in Children Depression Rating Scale - Revised (CDRS-R) Total Score at Week 26
Description: CDRS-R consisted of 17 items out of which 3 items rated nonverbal observations (listless speech, hypoactivity, and depressed affect). Fourteen items were rated on a 7-point scale from 1 to 7, and 3 items (sleep disturbance, appetite disturbance, and listless speech) were scored on a 5-point scale from 1 to 5. A rating of 1 indicated normal functioning and a higher number indicated a greater degree of depression. Total score ranged from 17 (normal) to 113 (severe depression). Least square (LS) mean was calculated using a restricted maximum likelihood-based mixed model for repeated measurements (MMRM) approach.
Time Frame: Baseline, Week 26
Population: Full analysis set (FAS) included all participants who took at least 1 dose of vortioxetine in this study 12712A with valid open-label extension baseline (OLEXA) assessment and at least 1 valid post-OLEXA assessment of the CDRS-R total score. Here, 'overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine
Number analyzed (Participants) | 506
units on a scale | -16.05 (0.63) [lower limit 0.63]

3. Secondary Outcome: Time to First Relapse
Description: Relapse was defined as a total score ≥40 on the CDRS-R. CDRS-R consisted of 17 items out of which 3 items rated nonverbal observations (listless speech, hypoactivity, and depressed affect). Fourteen items were rated on a 7-point scale from 1 to 7, and 3 items (sleep disturbance, appetite disturbance, and listless speech) were scored on a 5-point scale from 1 to 5. A rating of 1 indicated normal functioning and a higher number indicated a greater degree of depression. Total score ranged from 17 (normal) to 113 (severe depression).
Time Frame: Baseline up to Week 26
Population: Due to change in planned analysis, this endpoint was not analyzed; hence, data were not collected for this outcome measure.
Arm/Group | Vortioxetine
Number analyzed (Participants) | 0

4. Secondary Outcome: Time to First Loss of Remission
Description: Remission was defined as a total score ≤28 on the CDRS-R. CDRS-R consisted of 17 items out of which 3 items rated nonverbal observations (listless speech, hypoactivity, and depressed affect). Fourteen items were rated on a 7-point scale from 1 to 7, and 3 items (sleep disturbance, appetite disturbance, and listless speech) were scored on a 5-point scale from 1 to 5. A rating of 1 indicated normal functioning and a higher number indicated a greater degree of depression. Total score ranged from 17 (normal) to 113 (severe depression).
Time Frame: Baseline up to Week 26
Population: as for outcome 3
Arm/Group | Vortioxetine
Number analyzed (Participants) | 0

5. Secondary Outcome: Change From Baseline in Clinical Global Impression - Severity of Illness (CGI-S) Score at Week 26
Description: The CGI-S provides the clinician's impression of the participant's current state of mental illness. The clinician uses his or her clinical experience of this participant population to rate the severity of the participant's current mental illness on a 7-point scale ranging from 1 (normal - not at all ill) to 7 (among the most extremely ill participants). LS mean was calculated using a restricted maximum likelihood-based MMRM approach.
Time Frame: Baseline, Week 26
Population: FAS included all participants who took at least 1 dose of vortioxetine in this study 12712A with valid OLEXA assessment and at least 1 valid post-OLEXA assessment of the CDRS-R total score. Here, 'overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine
Number analyzed (Participants) | 506
units on a scale | -1.48 (0.06) [lower limit 0.06]

6. Secondary Outcome: Clinical Global Impression - Global Improvement (CGI-I) Score
Description: The CGI-I provides the clinician's impression of the participant's improvement (or worsening). The clinician assesses the participant's condition relative to a baseline on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). LS mean was calculated using a restricted maximum likelihood-based MMRM approach.
Time Frame: Week 26
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine
Number analyzed (Participants) | 506
units on a scale | 1.72 (0.04) [lower limit 0.04]

7. Secondary Outcome: Children (7-11 Years): Change From Baseline in Behaviour Rating Inventory of Executive Function - Preschool (BRIEF-P) Using the Global Executive Composite (GEC) Score at Week 26
Description: BRIEF form is an 86-item measure with symptoms rated on a 3-point likert scale of 1 "never", 2 "sometimes" or 3 "often". These items cover 8 non-overlapping clinical scales. For BRIEF-P form, only the first 72 items (Inhibit [10], Shift [8], Emotional Control [10], Initiate [8], Working Memory [10], Plan/Organize [12], Organization of Materials [6], Monitor [8]) were included in clinical scales. Clinical scales combined to form 2 indexes, Behavioural Regulation Index (BRI) and Metacognition Index (MI), and 1 composite summary score, the GEC, that incorporates all 8 clinical scales. GEC score was calculated as the sum of index scores ranging from 72-216; higher scores indicating greater impairment in executive functions. Raw scores converted to T-scores as detailed in T-score conversion tables for BRIEF-P. Conversion was based on gender and age group. T-scores ranged between 30 to 101, with a lower score indicating better functioning.
Time Frame: Baseline, Week 26
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Vortioxetine
Number analyzed (Participants) | 217
T score | -7.41 (11.70) [lower limit 11.70]

8. Secondary Outcome: Adolescents (12-18 Years): Change From Baseline in Behaviour Rating Inventory of Executive Function - Self-report (BRIEF-SR) Using the GEC Score at Week 26
Description: BRIEF form is an 86-item measure that assesses impairment in executive function with symptoms rated on a 3-point likert scale of 1 "never", 2 "sometimes" or 3 "often". These items cover 8 non-overlapping clinical scales. For BRIEF-SR form, only 80 items (Inhibit [13], Shift [10], Emotional Control [10], Initiate [5], Working Memory [12], Plan/Organize [13], Organization of Materials [7], Monitor [10]) were included in clinical scales. Clinical scales combined to form 2 indexes, the BRI and the MI, and 1 composite summary score, the GEC, that incorporates all 8 clinical scales. GEC score was calculated as the sum of index scores and ranges from 80-240 with higher scores indicating greater impairment in functions. Raw scores converted to T-scores as detailed in T-score conversion tables for BRIEF-SR. The conversion was based on gender and the age group. T-scores ranged between 29 to 104, with a lower score indicating better functioning.
Time Frame: Baseline, Week 26
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Vortioxetine
Number analyzed (Participants) | 272
T score | -7.50 (13.82) [lower limit 13.82]

9. Secondary Outcome: Children (7-11 Years): Change From Baseline in BRIEF-P Using the MI Score at Week 26
Description: BRIEF form is an 86-item measure that assesses impairment in executive function with symptoms rated on a 3-point likert scale of 1 "never", 2 "sometimes" or 3 "often". These items cover 8 non-overlapping clinical scales. Clinical scales combined to form 2 indexes, the BRI and the MI. For BRIEF-P, MI is comprised of Initiate (8), Working Memory (10), Plan/Organize (12), Organization of Materials (6), and Monitor (8) scales. The MI scores are calculated as the sum of the total 44 items ranging from 44 to 132 with lower scores reflecting better functioning. Raw scores converted to T-scores as detailed in T-score conversion tables for BRIEF-P. The conversion was based on gender and the age group. T-scores ranged between 30 to 98, with a lower score indicating better functioning.
Time Frame: Baseline, Week 26
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Vortioxetine
Number analyzed (Participants) | 217
T score | -7.36 (11.98) [lower limit 11.98]

10. Secondary Outcome: Adolescents (12-18 Years): Change From Baseline in BRIEF-SR Using the MI Score at Week 26
Description: BRIEF form is an 86-item measure that assesses impairment in executive function with symptoms rated on a 3-point likert scale of 1 "never", 2 "sometimes" or 3 "often". These items cover 8 non-overlapping clinical scales. Clinical scales combined to form 2 indexes, the BRI and the MI. For BRIEF-SR, MI is comprised of Working Memory (12), Plan/Organize (13), Organization of Materials (7), and Task Completion (10) scales. The MI scores are calculated as the sum of the total 42 items ranging from 42 to 126 with lower scores reflecting better functioning. Raw scores converted to T-scores as detailed in T-score conversion tables for BRIEF-SR. The conversion was based on gender and the age group. T-scores ranged between 31 to 100, with a lower score indicating better functioning.
Time Frame: Baseline, Week 26
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Vortioxetine
Number analyzed (Participants) | 272
T score | -7.18 (13.71) [lower limit 13.71]

11. Secondary Outcome: Change From Baseline in Children's Global Assessment Scale (CGAS) Score at Week 26
Description: The CGAS is a clinician-rated global scale to measure the lowest level of functioning for a child (4 to 16 years) during a specified time period. The CGAS contains behaviourally-oriented descriptors at each anchor point that depict behaviours and life situations applicable to a child. The score ranges from 1 (most functionally impaired child) to 100 (the healthiest). A score greater than 70 indicates normal function.
Time Frame: Baseline, Week 26
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vortioxetine
Number analyzed (Participants) | 506
units on a scale | 14.78 (14.29) [lower limit 14.29]

12. Secondary Outcome: Change From Baseline in Pediatric Quality of Life Inventory Present Functioning Visual Analogue Scale (PedsQL VAS) Total Score at Week 26
Description: The PedsQL™ VAS is designed to measure at-that-moment functioning in children and adolescents. The PedsQL™ VAS consists of 6 domains: anxiety, sadness, anger, worry, fatigue, and pain using VAS. The functionality for each domain is measured on a 10 cm line with a happy face at one end and a sad face at the other (0-10 points). The participants are asked to mark on the line how they feel. The total score is the average of all 6 items ranging from 0 to 10, where a lower value represents a better outcome.
Time Frame: Baseline, Week 26
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vortioxetine
Number analyzed (Participants) | 505
units on a scale | -1.50 (1.87) [lower limit 1.87]

13. Secondary Outcome: Number of Participants With Response to the Palatability Questionnaire
Description: The palatability of vortioxetine oral drops was assessed after intake of a single dose (5 to 20 mg) corresponding to the participant's current vortioxetine dose (replacing the vortioxetine tablet on that day). The palatability assessment included 4 questions on the overall appreciation of a medicinal product in relation to its taste (What do you think of the taste), mouthfeel (How does medicine feel in your mouth), aftertaste (What do you think of the after taste), and smell (What do you think of the smell). The items were rated on a 5-point hedonic scale; really bad, bad, neither good or bad, good, or very good. The oral drops were considered acceptable if the mean hedonic scores were ≤3 for each aspect of palatability (taste, aftertaste, smell, and mouthfeel).
Time Frame: assessed at Baseline up to Week 26, Week 26 reported
Population: APTS included all participants who took at least 1 dose of vortioxetine in this study 12712A. Here, 'overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Vortioxetine
Number analyzed (Participants) | 153
Participants
  Mouthfeel: Really bad | 11
  Mouthfeel: Bad | 17
  Mouthfeel: Neither good or bad | 38
  Mouthfeel: Good | 55
  Mouthfeel: Very good | 32
  Aftertaste: Really bad | 13
  Aftertaste: Bad | 26
  Aftertaste: Neither good or bad | 54
  Aftertaste: Good | 32
  Aftertaste: Very good | 28
  Smell: Really bad | 4
  Smell: Bad | 4
  Smell: Neither good or bad | 37
  Smell: Good | 59
  Smell: Very good | 49
  Taste: Really bad | 13
  Taste: Bad | 15
  Taste: Neither good or bad | 33
  Taste: Good | 60
  Taste: Very good | 32

14. Secondary Outcome: Number of Participants With Response to the Acceptability Questionnaire
Description: The acceptability of vortioxetine oral drops was assessed after intake of a single dose (5 to 20 mg) corresponding to the participant's current vortioxetine dose (replacing the vortioxetine tablet on that day). The acceptability assessment was based on 3 items; acceptability of the taste, whether the drops were perceived as easy to take, willingness to take the drops every day (provided it was the only available formulation). For each item the response options were no, not sure, and yes. The oral drops were considered acceptable if <60% of participants responded "no" to each of the 3 questions regarding acceptability.
Time Frame: assessed at Baseline up to Week 26, Week 26 reported
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | Vortioxetine
Number analyzed (Participants) | 153
participants
  Willingness to take the drops every day: No | 27
  Willingness to take the drops every day: Not sure | 17
  Willingness to take the drops every day: Yes | 109
  Easy to take medicine: No | 8
  Easy to take medicine: Neither easy or difficult | 10
  Easy to take medicine: Yes | 135
  Acceptability of the taste: No | 31
  Acceptability of the taste: Not sure | 24
  Acceptability of the taste: Yes | 98

ADVERSE EVENTS:
Time Frame: Baseline up to Week 30
Description: APTS included all participants who took at least 1 dose of vortioxetine in this study 12712A.
Arm/Group | Vortioxetine
All-Cause Mortality (participants affected / at risk) | 0/662
Serious Adverse Events (participants affected / at risk) | 14/662
Other Adverse Events (participants affected / at risk) | 255/662
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vortioxetine (N=662)
Intentional overdose (Injury, poisoning and procedural complications) | 3 (4)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (2)
Osteitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Torticollis (Musculoskeletal and connective tissue disorders) | 1 (1)
Psychomotor hyperactivity (Nervous system disorders) | 1 (1)
Major depression (Psychiatric disorders) | 1 (4)
Mania (Psychiatric disorders) | 1 (2)
Psychogenic seizure (Psychiatric disorders) | 1 (1)
Suicidal behaviour (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 4 (5)
Suicide attempt (Psychiatric disorders) | 4 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vortioxetine (N=662)
Abdominal pain (Gastrointestinal disorders) | 46 (58)
Nausea (Gastrointestinal disorders) | 138 (212)
Vomiting (Gastrointestinal disorders) | 69 (100)
Nasopharyngitis (Infections and infestations) | 46 (61)
Dizziness (Nervous system disorders) | 38 (55)
Headache (Nervous system disorders) | 116 (198)

LIMITATIONS AND CAVEATS:
The study was terminated early based on new efficacy data from another study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-01-16): https://cdn.clinicaltrials.gov/large-docs/97/NCT02871297/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/97/NCT02871297/SAP_001.pdf